CLINICAL TRIAL: NCT04543058
Title: Randomized Controlled Study of the Effectiveness of a Self-education Program When Walking by Rhythmic Auditory Stimulation Adapted Music, Delivered by BeatPark, in People With Parkinson's Disease
Brief Title: BeatPark: Self-rehabilitation in Walking With Parkinson's Disease
Acronym: BeatPark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Beau Soleil (Other)
Collaborators: Team Languedoc Mutualité / Nouvelles technologies (Unknown); University Hospital, Montpellier (Other); Euromov, Montpellier Univeristy (Unknown); Université de Montréal (Other); AxLR SATT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-A02032-55
Record Dates: First submitted 2020-07-06; First posted 2020-09-09 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Walking, Difficulty
Keywords: Walking rehabilitation; Parkinson Disease; Music
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BeatPark Experimental Group (Experimental): Group of participants who will make its self-rehabilitation in walking program using BeatPark application, delivering synchronized music adapted to the patient walking progression.
  Interventions: Device: BeatPark Application
- Control Group with Music at Random Tempo (Active Comparator): Group of participants who will make its self-rehabilitation in walking program using an application delivering music at random tempo.
  Interventions: Other: BeatPark Application without synchronized music
- Control Group without Music (Active Comparator): Group of participants who will make its self-rehabilitation in walking program using an application without music.
  Interventions: Other: BeatPark Application without music

INTERVENTIONS:
Device: BeatPark Application — The participant walks for 30 minutes a day, 5 day a week for 4 weeks. During the walking session, BeatPark Application delivers synchronized music adapted to the patient walking.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: BeatPark Experimental Group
Other: BeatPark Application without synchronized music — The participant walks for 30 minutes a day, 5 days a week for 4 weeks. During the walking session, BeatPark Application delivers random music at random tempo.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: Control Group with Music at Random Tempo
Other: BeatPark Application without music — The participant walks for 30 minutes a day, 5 days a week for 4 weeks. During the walking session, BeatPark Application does not deliver music. The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: Control Group without Music

SUMMARY:
Physical activity has beneficial effects on the quality of walking for persons with Parkinson's disease (PD). However, regular physical activity is still limited in most patients' daily lives.

The rhythm of music makes you want to move whether you are sick or not. In addition, it has been found that in people with PD, it can also improve walking by helping the participant to regain the regularity of alternating steps and a better walking dynamic (i.e. better position, better arm swinging, etc.). Studies have shown that music allows persons with PD to walk faster, with bigger steps.

However, if the tempo of the music does not correspond to the participant's walking pace, instead of helping him, it can disturb him. So it seems necessary for music to help people with PD to walk better if the tempo of the music is set to match their steps.

BeatPark is a smartphone application which makes it possible to synchronize the tempo of the music with the participant's walking rhythm detected thanks to feet insoles. Once synchronized to the participant's walking pace, BeatPark imperceptibly accelerates the tempo of the music to help the participant's acceleration.

This clinical trial proposes to study the effects of walking rehabilitation depending on the use of music synchronized to the participant's step with BeatPark, music with random tempo or without music.

DETAILED DESCRIPTION:
Groups, with and without music, will have the same visits and the same instructions throughout the study.

1. Visit 0 (inclusion visit)

   * Verification of inclusion and non-inclusion criteria
   * Signature of consent
   * Information gathering

     * Demographic information (date of birth, height, weight, activity, etc.) professional).
     * Clinical information about the disease (age of onset and duration of the disease, treatments and their distribution).
     * Medical history including present or past medical conditions and any other conditions that may be relevant to the study and their treatment.
   * Neurological examination with MDS-UPDRS (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) and NFOG-Q (New Freezing of Gait-Questionnaire) scales
   * Explanation and delivery of the agenda for the next 2 weeks
   * "Feetme(c)" soles in place
   * Remittance of self-questionnaires for a home refill before V1
2. Base Line From the day of inclusion until visit 1 the patient will complete a diary to record the occurrence of falls and freezing, and to self-assess on a visual numerical scale their levels of pain, fatigue and motivation.
3. Visit 1 (week 2)

   * Run the 6 minutes test in silence.
   * Actualization of the Battery for the Assessment of Auditory Sensorimotor and Timing Abilities (BAASTA).
   * Collecting and checking the completeness of the different scales given at visit 0 and helping to fill in incomplete scales.
   * Information and training in the use of the BeatPark device (programmed with or without music according to randomization)
   * Explanation of the self-education program (number of sessions, duration, location...) for the 4 weeks.
   * Delivery of questionnaires to be completed within 3 days prior to the visit 2.
   * MRI: morphological sequences (T1 3D, T2 FLAIR, T2*) and functional sequences (Resting state and with the different types of auditory indication) for the subgroup explored in imaging.
4. Intervention phase

   *Self-reeducation program:
   * This program will consist of walking outdoors for 5 sessions of 30 minutes per week for 4 consecutive weeks with the BeatPark device (set to deliver music or not, adapted music or random tempo).

     * Phone call:
   * The clinical research associate (CRA) will contact the patient to ensure the proper functioning and compliance with the rehabilitation program, if any difficulties are encountered.

     *Self-assessment schedule:
   * From the day of visit 1 through visit 2 the participant will complete a diary to record the occurrence of falls and freezing, and to self-assess on a visual numerical scale their levels of pain, fatigue, motivation and satisfaction.
5. Visit 2 (end-of-study visit, week 4):

   * Neurological evaluation with the MDS-UPDRS, NFOG and CGI (Clinical Global Impression) scales.
   * Running the 6 minutes test in silence
   * Achievement of the BAASTA
   * Collection and verification of the completeness of the different scales submitted to V1 (and completed within the last 3 days) and helps to fill in incomplete scales
   * Checking for no change in anti-parkinsonian treatment.
   * Return the equipment to the investigation team.
   * MRI: morphological sequences (T1 3D, T2 FLAIR, T2*) and functional sequences (Resting, T2 FLAIR, T2*). state and with the different types of auditory indication))) for the subgroup explored in imagery.

ELIGIBILITY:
Inclusion Criteria:

Specific Inclusion Criteria:

* Have a diagnosis of idiopathic PD according to the MDS clinical Diagnostic Criteria for PD (Postuma et al. 2015);
* Have a walking disorder defined by the neurologist (Item 10 of the MDSUPDRS-III ≥1);
* Be able to walk 30 consecutive minutes without technical assistance (e.g. cane or walker) or human assistance;
* Receive an uninterrupted antiparkinsonian pharmacological treatment since one month (and throughout the study period).

Non-Specific Inclusion Criteria:

* Be over 35 and under 95 of age;
* Be able to understand the nature, purpose and methodology of the study and agree to cooperate during assessments;
* Have signed the informed consent;
* Be affiliated to a social security plan or affiliated to such a equivalent health plan.

Non-Inclusions:

Specific Non-Inclusion Criteria:

* Presence of signs in favor of an atypical parkinsonian syndrome (involvement oculomotor, early falls, hallucinations, Montreal Cognitive Assessment <21/30, severe and early dysautonomia);
* Have a hearing impairment;
* Have any other neurological damage that affects walking;
* Have a walking disorder of other origin (e.g. orthopedic, rheumatological, etc.);
* Have severe or unbalanced heart or respiratory Failure which contraindicates walk rehabilitation.

Non-Specific Non-Inclusion Criteria:

* Adult under legal protection or unfit to express their consent (Article 1121-8 of the CSP);
* Vulnerable people (Article L 1121-6 of the CSP);
* Loss of liberty by judicial or administrative decision;
* High probability of non-compliance with the protocol or abandonment during the study;
* Pregnant / lactating women.

Non-Inclusion Criteria for the subgroup that will carry out the MRI ancillary study:

* Pacemaker or neurosensory stimulator or implantable defibrillator;
* Cochlear implants;
* Foreign ferromagnetic ocular or cerebral bodies close to nervous structures
* Metal prosthesis;
* Agitation of the participants: non-cooperative or agitated participants;
* Claustrophobic participants;
* Pregnant woman;
* Ventriculo-peritoneal neurosurgical bypass valves;
* Braces.

Exclusion Criteria:

* Participant no longer wishing to participate in the study, or during the study with refusal to use data until the time of the study exit;
* A change in the background treatment of PD will not systematically justify leaving the study but will be evaluated by the scientific committee on a case-by-case basis.

Ages: 36 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in average speeds | Up to 6 weeks
  The main outcome measure is the difference in average speeds measured during walking with musical stimulation during the last 10 minutes of the last 3 self-rehabilitation sessions.
  These speeds will be measured by the "Feetme(c)" soles under the same conditions ecological.
  If the subject stops his program before having completed the 20 full sessions, the speed will be evaluated over the last 3 fully completed rehabilitation sessions. Statistical analysis will be done with intent to treat. This criterion will be applied in main judgment to compare groups with music adapted and music at random tempo.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Cohen, M.D., Principal Investigator — Clinique Beau Soleil
Locations (1):
- Clinique Beau Soleil, Montpellier, Hérault, France